CLINICAL TRIAL: NCT03528512
Title: Comparison of Sedation, Pain, and Care Provider Satisfaction Between the Use of Intranasal Ketamine Versus Intranasal Midazolam and Fentanyl During Laceration Repair
Brief Title: IN Ketamine vs IN Midazolam and Fentanyl for Laceration Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Staffing for study was eliminated
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Margaret J Menoch, MD, Pediatric ER Medical Clinical Faculty, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-363
Record Dates: First submitted 2018-05-05; First posted 2018-05-18 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Laceration of Skin
Keywords: Pediatric; analgesia; pain control; sedation; intranasal ketamine; intranasal midazolam; intranasal fentanyl
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Midazolam; Fentanyl

STUDY DESIGN:
Intervention Model Description: Randomized double blinded control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization list created by an online randomization tool will be used to assign participants to a treatment arm (in random blocks of 4, 6, and 8). As participants are enrolled in the study, they will be assigned to the next available sequential treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IN ketamine (Experimental): Intranasal ketamine 3mg/kg (max 100 mg) + saline 0.03 ml/kg (max 2ml)
  Interventions: Drug: Ketamine
- IN midazolam and fentanyl (Active Comparator): Intranasal midazolam 0.3 mg/kg (max 10 mg) + fentanyl 1.5mcg/kg (max 100 mcg)
  Interventions: Drug: Midazolam and fentanyl

INTERVENTIONS:
Drug: Ketamine — Intranasal ketamine 3mg/kg (max 100 mg) + saline 0.03 ml/kg (max 2ml)
  Arms: IN ketamine
Drug: Midazolam and fentanyl — Intranasal midazolam 0.3 mg/kg (max 10 mg) + fentanyl 1.5mcg/kg (max 100 mcg)
  Arms: IN midazolam and fentanyl

SUMMARY:
Often, repair of the cuts (laceration repair) proves to be traumatic for the children and the parents. Nasal spray (Intranasal/IN) approaches for procedural pain reduction, such as during dental work, have been demonstrated to make drug administration painless and well tolerated. We are comparing IN ketamine to IN midazolam and fentanyl for pain and reducing anxiety during repair of cuts in children.

DETAILED DESCRIPTION:
Children frequently present to pediatric emergency center (PEC) with cuts of different body parts. Often, repair of the cuts (laceration repair) proves to be traumatic for the children and the parents alike. Ideally, repair of the cuts should be as painless and free from anxiety as possible. To work towards this goal, different analgesic (pain drugs) and sedative ( to calm patients down) management strategies use intravenous (into the vein), intramuscular ( into the muscle) and, more recently, intranasal (into the nostrils) routes. Unfortunately, intravenous access is hard to establish and may be painful for the child. The intramuscular route is often similarly painful. Due to the rich blood supply and large surface area of the nasal vestibule, intranasally (IN) administered medications are highly absorbed. IN approaches for procedural pain reduction, such as during dental work, have been demonstrated to make drug administration painless and well tolerated, making it an attractive potential alternative to commonly used intravenous and intramuscular approaches. In several small research studies, high doses of intranasal ketamine (9 mg/kg) produce adequate sedation during laceration repair with minimal side effects. A recent study compared IN ketamine, midazolam, fentanyl or combination of these drugs for pain management and urgent analgesia sedation, and demonstrated that they are effective and safe, reporting that ~60% of study participants sustained mild to moderate sedation. Unfortunately, there are not enough studies done to evaluate the sedation effect of IN ketamine for laceration repair. Small studies (Tsze and Nemeth) showed that IN ketamine is an effective alternative but no studies are done to compare combination IN midazolam and fentanyl to IN ketamine. Our null hypothesis is that there is no difference in sedation scores during laceration repair when comparing the use of IN ketamine to IN midazolam and IN fentanyl.

We will recruit a total of 30 pediatric patients (6 months - 10 y age) in a randomized double-blinded pilot study of IN ketamine alone or combined IN midazolam and IN fentanyl for laceration repair, comparing levels of pain and sedation scores using validated pediatric metrics as the primary outcomes. In addition, we will assess comparative nurse and physician satisfaction in each of these two groups. Understanding the relative effectiveness of these two approaches will help us identify a safe, effective, and easily administrable method to manage pain and anxiety, thereby, improving patient experience and outcomes during the often traumatic laceration repair procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 6 months to 10 years who required laceration repair in the pediatric emergency center.
* Laceration should be less than 5 cm long, require 2 or more sutures and no consult subspeciality consult for repair.
* Topical anesthetic (lidocaine-epinephrine-tetracaine topical solution/XAP) will be applied to all lacerations for 20 minutes duration before giving the intranasal medications.

Exclusion Criteria:

* Age < 6 months
* Documented allergy or adverse effect to ketamine, midazolam or fentanyl
* Epistaxis
* Partial upper airway obstruction
* Oxygen requirement via nasal cannula
* Acute mental status changes (e.g. obtunded or somnolent)
* Documented increased intracranial pressure or increased ocular pressure
* Documented porphyria
* Previously involved in the study
* Parent or patient refusal
* Acutely compromised vitals (hypotension, desaturations, respiratory distress)
* Any known heart disease
* If any previous opioid use for analgesia during the visit
* Need for staples
* Scalp wounds
* General trauma requiring additional sedation
* Patients who received pain medications (acetaminophen or ibuprofen) before laceration repair

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Levasseur, DO, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospital - Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IN Ketamine | IN Midazolam and Fentanyl
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IN Ketamine | IN Midazolam and Fentanyl | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 2 (0.87) | 2 (0) | 2 (0.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Sedation Score
Description: The primary outcome variable is the maximum sedation score as measured by the University of Michigan Sedation Scale. This scale consists of an ordinal scale from 0 being awake and alert and 4 being unarousable. Medians will be calculated for each group.
Time Frame: up to 30 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IN Ketamine | IN Midazolam and Fentanyl
Number analyzed (Participants) | 3 | 2
units on a scale | 1 [.5 to 1] | 1 [1 to 1]

2. Primary Outcome: Proportion of Children With Maximum Sedation Score
Description: The proportion of children who receive a maximum sedation score of either 1 or 2 (without distinguishing between those values)
Time Frame: Up to 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | IN Ketamine | IN Midazolam and Fentanyl
Number analyzed (Participants) | 3 | 2
Participants | 2 | 2

3. Secondary Outcome: Pain Scores During Laceration Repair
Description: The effect of IN ketamine vs IN midazolam + IN fentanyl on pain scores during laceration repair using either Face, Legs, Activity, Cry, Consolability (FLACC) Scale or Faces Scale pain scale depending for patient age, each a Likert scale from 0 being no pain to 10 being worst pain, median scores for each group
Time Frame: Up to 30 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IN Ketamine | IN Midazolam and Fentanyl
Number analyzed (Participants) | 3 | 2
units on a scale | 4 [4 to 4.5] | 0 [0 to 0]

4. Secondary Outcome: Nurse and Physician Satisfaction
Description: Nurse and physician satisfaction will be assessed by a survey which will be filled in the end of the sedation. Response to overall experience question score on Likert scale where 1 is poor and 5 is Excellent. Proportion of responders giving answers of 4 or 5 will be calculated.
Time Frame: Up to 30 minutes
Population: Two provider surveys were available for each patient experience
Measure: Count of Participants; unit: Participants
Arm/Group | IN Ketamine | IN Midazolam and Fentanyl
Number analyzed (Participants) | 6 | 4
Participants | 1 | 4

5. Secondary Outcome: Rates of Failure
Description: Rates of failure to repair laceration due to agitation or intolerable pain with the switch to intravenous medications will be compared between two groups. Percentage failure will be reported.
Time Frame: Up to 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | IN Ketamine | IN Midazolam and Fentanyl
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

6. Secondary Outcome: Change in Vitals
Description: Proportion of children who have any significant change in vitals during analgosedation (any desaturation - Oxygen saturation < 90, and hypotension per age-related norms) will be compared between the two groups.
Time Frame: up to 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | IN Ketamine | IN Midazolam and Fentanyl
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30-45 minutes
Arm/Group | IN Ketamine | IN Midazolam and Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

LIMITATIONS AND CAVEATS:
Study terminated early because staffing was eliminated. No results analyzed due to population size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03528512/Prot_SAP_001.pdf